CLINICAL TRIAL: NCT06418100
Title: Recto-intercostal Fascial Plane Block for Postoperative Analgesia in Coronary Artery Bypass Grafting With Sternotomy: a Randomized, Double-blind, Controlled Study
Brief Title: Recto-intercostal Block for Coronary Artery Bypass Grafting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 272-2023
Record Dates: First submitted 2024-02-26; First posted 2024-05-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease; Peripheral Nerve Blocks; Sternotomy
Keywords: coronary artery bypass grafting; Parasternal intercostal plane block; Recto-intercostal fascial plane block; Postoperative analgesia
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: prospective, randomized, triple-blind, controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants under general anaesthesia and the cardiovascular surgeon responsible for the study were blinded to the study groups. This surgeon served as the sole evaluator of postoperative outcomes. Intraoperative results were recorded by the anaesthesia technician, who was present in the operating room and unaware of the block procedures performed. Moreover, the data analysis was conducted before the unblinding of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Control (No Intervention): The participants will have standardized anaesthesia management and receive postoperative rescue analgesia as morphine.
- The rectointercostal fascial plane block (Experimental): The participants will receive postoperative recto intercostal fascial plane block, with 20 ml 0,25 bupivacaine bilaterally.
  Interventions: Procedure: The recto intercostal fascial plane block

INTERVENTIONS:
Procedure: The recto intercostal fascial plane block — After ensuring aseptic conditions, the high-frequency linear ultrasound probe was used to detect the rectus abdominis muscle and the 6-7th costal cartilage as described by Tulgar et al. After rotating and shifting the transducer, 6-7th costal cartilages, the rectus abdominis muscle, and intercostal muscles between the cartilages were confirmed. The primary investigator (B.C.) directed the needle tip caudad in the cephalic direction in-plainly, and 20 ml 0,25% bupivacaine was injected bilaterally into the plane between the costal cartilage and the rectus abdominis muscle following negative aspiration.
  Arms: The rectointercostal fascial plane block

SUMMARY:
This interventional study aims to learn about the postoperative analgesic efficacy of a new fascial plane block, recto-intercostal fascial plane block, at coronary artery bypass grafting with sternotomy. There will be two groups, one of which will be the control group, and the other will be the study group randomly receiving postoperative recto-intercostal fascial plane block.

The main questions it aims to answer are the effect of this new block on postoperative opioid consumption and pain scores. Also, postoperative outcomes related to respiratory ( postoperative oxygenation and atelectasis score), hemodynamic functions ( newly developed arrhythmias), total postanesthesia care unit stay, and hospital stay will be questioned.

DETAILED DESCRIPTION:
All patients will receive standard general anaesthesia under standard monitoring along with the bispectral index (Medtronic). Intubation will be performed by administering intravenous (IV) 0,03 mg/kg midazolam, propofol (Lipuro, Braun, max. 2 mg/kg according to BIS), two mcg/kg fentanyl (Talinat, VEM), 1 mg /kg rocuronium (Esmeron, Alessandroorsini) followed by 1 MAC sevoflurane (Sevorane, Abbott) in an air-oxygen mixture for maintenance of anaesthesia. Following anaesthesia induction, all participants will receive superficial parasternal intercostal plane block (SPIP) bilaterally along with 8 mg dexamethasone before surgical incision as part of multimodal analgesia by a single experienced regional anaesthesiologist (B.C.) under ultrasound guidance (Esaote MyLab ™ Seven). SPIPB will be performed using a high-frequency probe to visualize the pectointercostal fascial area at the intercostal level of the intercostal 3-4 level, and 20 ml %0,25 bupivacaine was injected bilaterally. After applying SPIPB, the surgery is set to begin after at least 15 minutes of block procedure. The intraoperative analgesic need will be supplied by fentanyl bolus doses as 50 mcq if necessary, as heart rate or systolic blood pressure increases by more than %15. According to randomization, the intervention group will receive RIFPB with 10 ml %0,25 bupivacaine.

From the beginning of acclaimed arousal till the 24th hour, rescue analgesia as tramadol 100 mg (maximum daily dose 400 mg) is applied if NRS is over four or with the patient's request. The routine analgesia regimen was 1 gram IV paracetamol 6th hourly postoperatively at the PACU. All patients were followed up from the extubation time till hospital discharge to evaluate respiratory and hemodynamic changes, possible complications and total postoperative time.

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo CABG surgery with sternotomy
* patients who have an American Society of Anesthesiologists (ASA) Physical Status classification of III to IV

Exclusion Criteria:

* refusal to participate
* a history of neurological deficits or neuropathy affecting the thoracal innervation
* infection at the site of block application
* allergy to local anesthetics
* epilepsy or treatment with antipsychotics
* abuse of alcohol or drugs
* previous surgery distorting the anatomy of the sternum, thorax or upper abdominal area
* severe organ dysfunction ( kidney, liver and other); patients who fail at weaning after 12 hours of surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Total rescue analgesic | postoperative 24 hour
  . From the beginning of acclaimed arousal till the 24th hour, rescue analgesia as tramadol 100 mg (maximum daily dose 400 mg) is applied if NRS over 4 or with the patient's request.

SECONDARY OUTCOMES:
intraoperative opioid use | intraoperative
  total amount of opioid use as fentanyl intraoperatively
intraoperative hemodynamic change | at sternotomy
  systolic blood pressure
postoperative respiratory function | postoperative 48 hour
  postoperative atelectasis score
postoperative arythmias | postoperative 48 hour
  postoperative arythmias especially atrial fibrillation

OTHER OUTCOMES:
total hospital stay | postoperative
  up to discharge postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, Principal Investigator — Haseki Training and Research Hospital Anesthesiology and Reanimation Department
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Alver S, Sakul BU, Ansen G, Pence KB, Alici HA. Recto-intercostal fascial plane block: Another novel fascial plane block. J Clin Anesth. 2023 Oct;89:111163. doi: 10.1016/j.jclinane.2023.111163. Epub 2023 Jun 7. No abstract available. PMID 37295124
- [Background] Chen Y, Li Q, Liao Y, Wang X, Zhan MY, Li YY, Liu GJ, Xiao L. Preemptive deep parasternal intercostal plane block for perioperative analgesia in coronary artery bypass grafting with sternotomy: a randomized, observer-blind, controlled study. Ann Med. 2023;55(2):2302983. doi: 10.1080/07853890.2024.2302983. Epub 2024 Feb 20. PMID 38375661